CLINICAL TRIAL: NCT04420312
Title: Incidence and Characteristics of Pulmonary Embolism in COVID-19 Patients Hospitalized for Acute Respiratory Syndrome
Brief Title: Prevalence and Characteristics of Pulmonary Embolism on COVID-19 Patients Presenting Respiratory Symptoms
Acronym: COVID-EP
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-EP; MR 4516150520 (Other: INDS)
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Pulmonary Embolism; Covid-19
Keywords: pulmonary embolism; covid-19; CT; D-Dimers; ARDS
MeSH Terms: conditions — Pulmonary Embolism; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Group 1: Enrolled the Covid-19 patients with a negative CT Pulmonary Angiogram.
- Group 2: Enrolled the Covid-19 patients in whom only a CT was performed.

SUMMARY:
Multicentric case-control study that is aims at:

* evaluating the prevalence of pulmonary embolism among a large population of consecutive patients admitted for COVID-19 pneumonia into two large university hospitals in Paris, France: Groupe Hospitalier Paris Saint-Joseph (GHPSJ) and Hôpital Européen Georges Pompidou (HEGP)
* and identifying the characteristics associated with pulmonary embolism by using a nested case control study design within the patients who underwent either unenhanced computed tomograpghy (CT) or CT pulmonary angiogram (CTPA) evaluation.

DETAILED DESCRIPTION:
In December 2019, China reported the first cluster of severe acute respiratory syndrome due to a new coronavirus (SARS-CoV-2). The disease rapidly spread into a global pandemic of public health emergency worldwide leading to more than 330.000 deaths (data from May 25th, 2020). We have, to date, no demonstration on the efficacy of any drug to cure or prevent severe evolution of the disease (COVID-19). The primary target of SARS-CoV-2 is the lung with frequent occurrence of acute respiratory distress syndrome (ARDS) justifying supportive care, including invasive mechanical ventilation (IMV). The characteristics of ARDS in COVID-19 patients appeared atypical due to the dissociation between initial well-conserved lung compliance and severe hypoxemia, attributed to pulmonary vasoregulation disruption and local thrombogenesis. Strikingly high D-dimers levels, caused by both inflammation storm and coagulation activation, have been early reported in COVID-19 patients and have been associated with increased mortality. A single observational study suggests that anticoagulation is associated with a decreased mortality in severe COVID-19 patients. These reports have led to several therapeutic propositions in terms of anticoagulant therapy from worldwide scientific societies (Khider et al JMV 2020). Publications recently reported thrombotic complications in series of severe COVID-19 patients admitted in ICU, but the frequency of pulmonary embolism (PE) in larger cohort of COVID-19 patients of any severity remains uncertain.

This cohort enrolled patients in whom PE is proven by CTPA and compared them into two subgroups of controls matched for age and sex in whom PE was either excluded or non suspected:

1. COVID-19 patients with a negative CTPA and
2. COVID-19 patients in whom only an unhenced CT was performed.

ELIGIBILITY:
Inclusion Criteria:

* patients >18 years,
* admitted for acute COVID-19 pneumonia and have recieved a chest CT scan during hospitalization,
* COVID-19 diagnosis confirmed by a positive result of a RT-PCR,
* CT findings of COVID-19 pneumonia.

Exclusion Criteria:

* Respiratory distress syndrome explained by other cause
* Patients who refuse to participate to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged over 18 years, hospitalized for respiratory pathology, associated with the COVID-19; confirmed by either a RT-PCR test or a CT scan.
Sampling Method: Probability Sample
Enrollment: 1024 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Impact of PE on COVID-19 patients | March 1st, 2020
  Evaluate the prevalence of Pulmonary embolism among a large population of consecutive COVID-19 patients presenting respiratory symptoms

SECONDARY OUTCOMES:
Clinical and radiological characteristics | April 20th,2020
  Identify the clinical, radiological or biological characteristics associated with pulmonary embolism.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Baden LR, Rubin EJ. Covid-19 - The Search for Effective Therapy. N Engl J Med. 2020 May 7;382(19):1851-1852. doi: 10.1056/NEJMe2005477. Epub 2020 Mar 18. No abstract available. PMID 32187463
- [Background] Chen T, Wu D, Chen H, Yan W, Yang D, Chen G, Ma K, Xu D, Yu H, Wang H, Wang T, Guo W, Chen J, Ding C, Zhang X, Huang J, Han M, Li S, Luo X, Zhao J, Ning Q. Clinical characteristics of 113 deceased patients with coronavirus disease 2019: retrospective study. BMJ. 2020 Mar 26;368:m1091. doi: 10.1136/bmj.m1091. PMID 32217556
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Tang N, Li D, Wang X, Sun Z. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 Apr;18(4):844-847. doi: 10.1111/jth.14768. Epub 2020 Mar 13. PMID 32073213
- [Background] Han H, Yang L, Liu R, Liu F, Wu KL, Li J, Liu XH, Zhu CL. Prominent changes in blood coagulation of patients with SARS-CoV-2 infection. Clin Chem Lab Med. 2020 Jun 25;58(7):1116-1120. doi: 10.1515/cclm-2020-0188. PMID 32172226
- [Background] Tang N, Bai H, Chen X, Gong J, Li D, Sun Z. Anticoagulant treatment is associated with decreased mortality in severe coronavirus disease 2019 patients with coagulopathy. J Thromb Haemost. 2020 May;18(5):1094-1099. doi: 10.1111/jth.14817. Epub 2020 Apr 27. PMID 32220112
- [Background] Marietta M, Ageno W, Artoni A, De Candia E, Gresele P, Marchetti M, Marcucci R, Tripodi A. COVID-19 and haemostasis: a position paper from Italian Society on Thrombosis and Haemostasis (SISET). Blood Transfus. 2020 May;18(3):167-169. doi: 10.2450/2020.0083-20. Epub 2020 Apr 8. No abstract available. PMID 32281926
- [Background] Akima S, McLintock C, Hunt BJ. RE: ISTH interim guidance to recognition and management of coagulopathy in COVID-19. J Thromb Haemost. 2020 Aug;18(8):2057-2058. doi: 10.1111/jth.14853. Epub 2020 Jul 15. No abstract available. PMID 32302442
- [Background] Bikdeli B, Madhavan MV, Jimenez D, Chuich T, Dreyfus I, Driggin E, Nigoghossian C, Ageno W, Madjid M, Guo Y, Tang LV, Hu Y, Giri J, Cushman M, Quere I, Dimakakos EP, Gibson CM, Lippi G, Favaloro EJ, Fareed J, Caprini JA, Tafur AJ, Burton JR, Francese DP, Wang EY, Falanga A, McLintock C, Hunt BJ, Spyropoulos AC, Barnes GD, Eikelboom JW, Weinberg I, Schulman S, Carrier M, Piazza G, Beckman JA, Steg PG, Stone GW, Rosenkranz S, Goldhaber SZ, Parikh SA, Monreal M, Krumholz HM, Konstantinides SV, Weitz JI, Lip GYH; Global COVID-19 Thrombosis Collaborative Group, Endorsed by the ISTH, NATF, ESVM, and the IUA, Supported by the ESC Working Group on Pulmonary Circulation and Right Ventricular Function. COVID-19 and Thrombotic or Thromboembolic Disease: Implications for Prevention, Antithrombotic Therapy, and Follow-Up: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Jun 16;75(23):2950-2973. doi: 10.1016/j.jacc.2020.04.031. Epub 2020 Apr 17. PMID 32311448
- [Background] Oudkerk M, Buller HR, Kuijpers D, van Es N, Oudkerk SF, McLoud T, Gommers D, van Dissel J, Ten Cate H, van Beek EJR. Diagnosis, Prevention, and Treatment of Thromboembolic Complications in COVID-19: Report of the National Institute for Public Health of the Netherlands. Radiology. 2020 Oct;297(1):E216-E222. doi: 10.1148/radiol.2020201629. Epub 2020 Apr 23. PMID 32324101
- [Background] Leonard-Lorant I, Delabranche X, Severac F, Helms J, Pauzet C, Collange O, Schneider F, Labani A, Bilbault P, Moliere S, Leyendecker P, Roy C, Ohana M. Acute Pulmonary Embolism in Patients with COVID-19 at CT Angiography and Relationship to d-Dimer Levels. Radiology. 2020 Sep;296(3):E189-E191. doi: 10.1148/radiol.2020201561. Epub 2020 Apr 23. PMID 32324102
- [Background] Grillet F, Behr J, Calame P, Aubry S, Delabrousse E. Acute Pulmonary Embolism Associated with COVID-19 Pneumonia Detected with Pulmonary CT Angiography. Radiology. 2020 Sep;296(3):E186-E188. doi: 10.1148/radiol.2020201544. Epub 2020 Apr 23. PMID 32324103
- [Background] Poissy J, Goutay J, Caplan M, Parmentier E, Duburcq T, Lassalle F, Jeanpierre E, Rauch A, Labreuche J, Susen S; Lille ICU Haemostasis COVID-19 Group. Pulmonary Embolism in Patients With COVID-19: Awareness of an Increased Prevalence. Circulation. 2020 Jul 14;142(2):184-186. doi: 10.1161/CIRCULATIONAHA.120.047430. Epub 2020 Apr 24. No abstract available. PMID 32330083
- [Background] Klok FA, Kruip MJHA, van der Meer NJM, Arbous MS, Gommers DAMPJ, Kant KM, Kaptein FHJ, van Paassen J, Stals MAM, Huisman MV, Endeman H. Incidence of thrombotic complications in critically ill ICU patients with COVID-19. Thromb Res. 2020 Jul;191:145-147. doi: 10.1016/j.thromres.2020.04.013. Epub 2020 Apr 10. PMID 32291094
- [Background] Helms J, Tacquard C, Severac F, Leonard-Lorant I, Ohana M, Delabranche X, Merdji H, Clere-Jehl R, Schenck M, Fagot Gandet F, Fafi-Kremer S, Castelain V, Schneider F, Grunebaum L, Angles-Cano E, Sattler L, Mertes PM, Meziani F; CRICS TRIGGERSEP Group (Clinical Research in Intensive Care and Sepsis Trial Group for Global Evaluation and Research in Sepsis). High risk of thrombosis in patients with severe SARS-CoV-2 infection: a multicenter prospective cohort study. Intensive Care Med. 2020 Jun;46(6):1089-1098. doi: 10.1007/s00134-020-06062-x. Epub 2020 May 4. PMID 32367170
- [Background] Middeldorp S, Coppens M, van Haaps TF, Foppen M, Vlaar AP, Muller MCA, Bouman CCS, Beenen LFM, Kootte RS, Heijmans J, Smits LP, Bonta PI, van Es N. Incidence of venous thromboembolism in hospitalized patients with COVID-19. J Thromb Haemost. 2020 Aug;18(8):1995-2002. doi: 10.1111/jth.14888. Epub 2020 Jul 27. PMID 32369666
- [Background] Lodigiani C, Iapichino G, Carenzo L, Cecconi M, Ferrazzi P, Sebastian T, Kucher N, Studt JD, Sacco C, Bertuzzi A, Sandri MT, Barco S; Humanitas COVID-19 Task Force. Venous and arterial thromboembolic complications in COVID-19 patients admitted to an academic hospital in Milan, Italy. Thromb Res. 2020 Jul;191:9-14. doi: 10.1016/j.thromres.2020.04.024. Epub 2020 Apr 23. PMID 32353746
- [Background] Revel MP, Parkar AP, Prosch H, Silva M, Sverzellati N, Gleeson F, Brady A; European Society of Radiology (ESR) and the European Society of Thoracic Imaging (ESTI). COVID-19 patients and the radiology department - advice from the European Society of Radiology (ESR) and the European Society of Thoracic Imaging (ESTI). Eur Radiol. 2020 Sep;30(9):4903-4909. doi: 10.1007/s00330-020-06865-y. Epub 2020 Apr 20. PMID 32314058
- [Background] PROTECT Investigators for the Canadian Critical Care Trials Group and the Australian and New Zealand Intensive Care Society Clinical Trials Group; Cook D, Meade M, Guyatt G, Walter S, Heels-Ansdell D, Warkentin TE, Zytaruk N, Crowther M, Geerts W, Cooper DJ, Vallance S, Qushmaq I, Rocha M, Berwanger O, Vlahakis NE. Dalteparin versus unfractionated heparin in critically ill patients. N Engl J Med. 2011 Apr 7;364(14):1305-14. doi: 10.1056/NEJMoa1014475. Epub 2011 Mar 22. PMID 21417952
- [Background] Hull RD, Schellong SM, Tapson VF, Monreal M, Samama MM, Nicol P, Vicaut E, Turpie AG, Yusen RD; EXCLAIM (Extended Prophylaxis for Venous ThromboEmbolism in Acutely Ill Medical Patients With Prolonged Immobilization) study. Extended-duration venous thromboembolism prophylaxis in acutely ill medical patients with recently reduced mobility: a randomized trial. Ann Intern Med. 2010 Jul 6;153(1):8-18. doi: 10.7326/0003-4819-153-1-201007060-00004. PMID 20621900
- [Background] Goldhaber SZ, Leizorovicz A, Kakkar AK, Haas SK, Merli G, Knabb RM, Weitz JI; ADOPT Trial Investigators. Apixaban versus enoxaparin for thromboprophylaxis in medically ill patients. N Engl J Med. 2011 Dec 8;365(23):2167-77. doi: 10.1056/NEJMoa1110899. Epub 2011 Nov 13. PMID 22077144
- [Background] Cohen AT, Spiro TE, Buller HR, Haskell L, Hu D, Hull R, Mebazaa A, Merli G, Schellong S, Spyropoulos AC, Tapson V; MAGELLAN Investigators. Rivaroxaban for thromboprophylaxis in acutely ill medical patients. N Engl J Med. 2013 Feb 7;368(6):513-23. doi: 10.1056/NEJMoa1111096. PMID 23388003
- [Background] Cohen AT, Harrington RA, Goldhaber SZ, Hull RD, Wiens BL, Gold A, Hernandez AF, Gibson CM; APEX Investigators. Extended Thromboprophylaxis with Betrixaban in Acutely Ill Medical Patients. N Engl J Med. 2016 Aug 11;375(6):534-44. doi: 10.1056/NEJMoa1601747. Epub 2016 May 27. PMID 27232649